CLINICAL TRIAL: NCT06449677
Title: A Randomized Trial of the Insulin-only Bionic Pancreas in Cystic Fibrosis Related Diabetes
Brief Title: Bionic Pancreas in CFRD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Massachusetts General Hospital (Other); Beta Bionics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPCFRD
Record Dates: First submitted 2024-05-20; First posted 2024-06-10 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis-related Diabetes
Keywords: Cystic fibrosis-related diabetes (CFRD); iLet bionic pancreas; Automated insulin delivery; Continuous glucose monitoring

STUDY DESIGN:
Intervention Model Description: 13-week RCT followed by a 13-week Extension Phase in which all participants use the iLet BP System
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- UC Group (Active Comparator): Participants randomized to the Usual Care (UC) group will use their existing insulin delivery method in conjunction with a study CGM during the first 13-week of the study (RCT phase). The UC group will then initiate use of the BP System for the remaining 13 weeks of the study (Extension Phase).
  Interventions: Device: iLet Bionic Pancreas System (BP); Device: Usual Care (UC)
- BP Group (Experimental): Participants randomized to the intervention group will use the BP group using the iLet Bionic Pancreas System (BP) and continuous glucose monitoring (CGM) during the first 13-week of the study (RCT phase). After the RCT phase, participants will continue in a 13-week Extension Phase in which the BP group will continue to use the BP system.
  Interventions: Device: iLet Bionic Pancreas System (BP)

INTERVENTIONS:
Device: iLet Bionic Pancreas System (BP) — The iLet Bionic Pancreas System (BP) consists of an integrated infusion pump, touchscreen display, Bluetooth radio, and insulin dosing algorithms, that automatically controls insulin delivery based on glucose values obtained by communicating with a CGM sensor.
Device: Usual Care (UC) — Usual Care consists in the participant existing insulin therapy (prior to enrollment) in conjunction with a study CGM. Existing insulin therapies are defined as multiple daily injections of insulin (MDI) or use of an insulin pump.
  Arms: UC Group

SUMMARY:
This multi-center randomized controlled trial (RCT) will compare efficacy and safety endpoints using the insulin-only configuration of the iLet Bionic Pancreas System (BP) versus a control group using their usual care insulin delivery method and continuous glucose monitoring (CGM) during a 13-week study period in individuals ≥14 years old with cystic fibrosis-related diabetes (CFRD). After 13 weeks, participants will continue in a 13-week Extension Phase in which the BP group will continue to use the BP system and the Usual Care group will initiate use of the BP system.

ELIGIBILITY:
Inclusion

1. Age ≥ 14 years old at time of signing informed consent
2. Able to provide informed consent (and assent for participants <18 years old)
3. Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

   * Sweat chloride equal to or greater than 60 mmol/liter by quantitative pilocarpine iontophoresis test (QPIT) (when not taking a cystic fibrosis transmembrane conductance regulator (CFTR) modulator)
   * Two well-characterized mutations in the CFTR gene
4. Clinical diagnosis of CFRD, defined as a person with CF and diabetes mellitus, treated with insulin for ≥3 months prior to screening
5. Using the same insulin regimen for ≥1 month prior to screening and collection of baseline CGM data, with no plans to change regimen during the study: either multiple daily injections of insulin (MDI), basal-only without bolus insulin, an insulin pump without automation, or an automated insulin delivery (AID) system other than the BP (which is an exclusion)
6. Total daily insulin dose must be ≥0.1 units/kg
7. Able to speak and read English sufficient to understand the pump user interface and provide written materials for safe operation of the BP

   • For pediatric participants, this applies to both the participant and caregiver
8. For participants <18 years old, living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia. A designated care partner must be willing to be linked to the participant's Dexcom Follow application with location sharing on.
9. For participants >18 years old who live alone, participant has a relative or acquaintance who lives within 30 minutes of participant and is willing to be contacted to check on participant if study staff feel that participant may be experiencing a medical emergency and cannot be reached. A designated care partner must be willing to be linked to the participant's Dexcom Follow application with location sharing on.
10. No use of a non-insulin glucose-lowering medication, except metformin, that is not approved for use in T1D within 3 months prior to signing informed consent and willing to not use any such medications during the course of the trial. Note: such drugs cannot be used even if prescribed for weight loss rather than glucose-lowering.
11. If not currently using a rapid-acting insulin that is approved for use in the iLet pump, willing and able to switch to an approved insulin when using the BP.
12. Participant has commercial glucagon available for treatment of severe hypoglycemia or will obtain it prior to randomization
13. Willing to authorize the study team to contact the participant's primary physician to inform them about their participation in this study.
14. Enrolled in the Cystic Fibrosis Foundation Patient Registry (participants may enroll in the Registry at the time of enrollment if not already enrolled).
15. No plans for trips of more than 14 consecutive days outside the United States during the period of study participation
16. Investigator believes that the participant can safely use the iLet and will follow the protocol • The investigator will take into account the participant's HbA1c level (there is no upper limit for eligibility), compliance with current diabetes management, prior acute diabetic complications, cognitive ability, and general medical condition. For this reason, there is no upper limit on HbA1c specified for eligibility.

Exclusion

1. Current use of the BP or an AID system not FDA approved for T1D
2. Known hemoglobinopathy (sickle cell trait is not an exclusion)
3. Current participation in another diabetes-related interventional trial
4. Established history of allergy or severe reaction to adhesive or tape that must be used in the study
5. Pregnant (positive urine hCG), breast feeding, plan to become pregnant in the next 7 months, or sexually active and can become pregnant but not using contraception
6. Current use of hydroxyurea or unable to avoid hydroxyurea use during the study (interferes with accuracy of Dexcom sensor)
7. Have started or stopped a CFTR modulator in the 4 weeks prior to screening.

   • Modifications of the dosing of a CFTR modulator is acceptable
8. Anticipated lung or liver transplant (on transplant list)
9. Lung or liver transplant within one year prior to screening. If they have had a transplant more than a year ago, but they:

   * Have had a rejection episode occur in prior 8 weeks, individual is excluded.
   * Their doses of corticosteroids and/or calcineurin inhibitors have not been stable for one month prior to enrollment and/or is expected to change significantly over the course of the study, individual is excluded.
10. Acute pulmonary exacerbation or hospitalization within the 4 weeks prior to screening or treatment with IV antibiotics in the 4 weeks prior to screening
11. History of a complete pancreatectomy
12. Currently using enteral tube feedings for nutritional support
13. Presence of a medical condition or use of a medication that, in the judgment of the investigator, clinical protocol chair, or medical monitor, could compromise the results of the study or the safety of the participant. Conditions to be considered by the investigator may include the following:

    * Alcohol or drug abuse
    * Use of prescription drugs that may dull the sensorium, or hinder decision-making during the period of participation in the study such has opioids or short-acting benzodiazepines
    * Coronary artery disease that is not stable with medical management, including unstable angina, angina that prevents moderate exercise (e.g., climbing a flight of stairs) despite medical management; or within the last 12 months before screening: a history of myocardial infarction, percutaneous coronary intervention, enzymatic lysis of a presumed coronary occlusion, or coronary artery bypass grafting
    * Congestive heart failure with New York Heart Association (NYHA) Functional Classification III or IV
    * History of TIA or stroke in the last 12 months
    * Severe liver disease such as end-stage cirrhosis
    * Renal failure requiring dialysis or known eGFR <30
    * Untreated or inadequately treated mental illness
    * History of untreated or inadequately treated eating disorder within the last 2 years, such as anorexia, bulimia, or diabulimia or omission of insulin to manipulate weight
    * History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
14. Employed by, or having immediate family members employed by Beta Bionics, or being directly involved in conducting the clinical trial, or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
CGM-measured Time In Target Range of 70-180 mg/dL (TIR) | 13 weeks
  CGM-measured time in target range of 70-180 mg/dL (TIR)

SECONDARY OUTCOMES:
CGM-measured Time In Range <54 mg/dL | 13 weeks
  CGM-measured time in range <54 mg/dL

OTHER OUTCOMES:
CGM-measured Mean Glucose | 13 weeks
  Average glucose value measured by CGM
CGM-measured Time In Range >180 mg/dL | 13 weeks
  CGM-measured time in range >180 mg/dL
CGM-measured Time In Range >250 mg/dL | 13 weeks
  CGM-measured time in range >250 mg/dL
HbA1c At 13 Weeks | 13 weeks
  HbA1c at 13 weeks
Glucose Variability Measured With the Standard Deviation (SD) | 13 weeks
  Glucose variability measured with the standard deviation (SD)
CGM-measured Time In Range <70 mg/dL | 13 weeks
  CGM-measured time in range <70 mg/dL
Glucose Variability With the Coefficient of Variation (CV) | 13 weeks
  Glucose variability with the coefficient of variation (CV)
HbA1c <7.0% At 13 Weeks | 13 weeks
  HbA1c <7.0% at 13 weeks
HbA1c <7.0% At 13 Weeks In Participants With Baseline HbA1c >7.5% | 13 weeks
  HbA1c <7.0% at 13 weeks in participants with baseline HbA1c >7.5%
HbA1c <8.0% At 13 Weeks | 13 weeks
  HbA1c <8.0% at 13 weeks
HbA1c Improvement From Baseline To 13 Weeks >0.5% | 13 weeks
  HbA1c improvement from baseline to 13 weeks >0.5%
HbA1c Improvement From Baseline To 13 Weeks >1.0% | 13 weeks
  HbA1c improvement from baseline to 13 weeks >1.0%
HbA1c Improvement From Baseline To 13 Weeks >1.0% Or HbA1c <7.0% At 13 Weeks | 13 weeks
  HbA1c improvement from baseline to 13 weeks >1.0% or HbA1c <7.0% at 13 weeks
CGM-measured Time In Tight Range (TITR) 70-140 mg/dL | 13 weeks
  CGM-measured time in tight range (TITR) 70-140 mg/dL
CGM-measured Area Over the Curve (70 mg/dL) | 13 weeks
  CGM-measured area over the curve (70 mg/dL)
CGM-measured Low Sensor Glucose Events | 13 weeks
  CGM-measured low sensor glucose events
CGM-measured Prolonged High Sensor Glucose Events | 13 weeks
  CGM-measured prolonged high sensor glucose events
CGM-measured Time >300 mg/dL | 13 weeks
  CGM-measured time >300 mg/dL
CGM-measured Area Under the Curve (180 mg/dL) | 13 weeks
  CGM-measured area under the curve (180 mg/dL)
CGM-measured TIR >70% | 13 weeks
  CGM-measured TIR >70%
CGM-measured TIR Improvement From Baseline To 13 Weeks ≥5% | 13 weeks
  CGM-measured TIR improvement from baseline to 13 weeks ≥5%
CGM-measured TIR Improvement From Baseline To 13 Weeks ≥10% | 13 weeks
  CGM-measured TIR improvement from baseline to 13 weeks ≥10%
CGM-measured Time <70 mg/dL <4% | 13 weeks
  CGM-measured time <70 mg/dL <4%
CGM-measured Time <54 mg/dL <1% | 13 weeks
  CGM-measured time <54 mg/dL <1%
CGM-measured TIR >70% and Time <54 mg/dL <1% | 13 weeks
  CGM-measured TIR >70% and time <54 mg/dL <1%
CGM-measured Improvement In TIR By >10% Without An Increase In Time <54 mg/dL By >0.5% | 13 weeks
  CGM-measured improvement in TIR by >10% without an increase in time <54 mg/dL by >0.5%
Type 1 Diabetes Distress Scale (T1-DDS) | Screening, 13 weeks
  The T1-DDS is to evaluate diabetes-related emotional distress in type 1 diabetic patients. The scale consists of 17 items, contains 4 domains (emotional burden subscale, physician-related subscale, regimen-related distress subscale, and diabetes-related interpersonal distress). Each item is rated on a 6-point Likert scale from 1 (no problem) to 6 (serious problem). Patients with higher scores are considered with more distress
Problem Areas In Diabetes - Teens (PAID-T) and Parents of Teens (P-PAID-T) | Screening, 13 weeks
  The PAID-T and P-PAID-T questionnaires consist of 26 items that are scored on a 6-point Likert scale from 1-2 (not a problem) to 5-6 (serious problem). The derived total score (26 questions) ranges between 26 and 156, where high scores represent a higher burden
Hypoglycemia Confidence Scale (≥18) | Screening, 13 weeks
  A person-reported outcome measure (PROM) that examines the degree to which people with diabetes feel able, secure, and comfortable regarding their ability to stay safe from hypoglycemic-related problems (9-item scale with 4 choices that range from 1 (Not Confident At All) to 4 (Very Confident)). The total score can range from 1 to 4, with a higher score indicating a better outcome
INSPIRE Survey (Insulin Delivery Systems: Perceptions, Ideas, Reflections, and Expectations) | Screening, 13 weeks
  INSPIRE 5-point Likert scale from strongly agree to strongly disagree, along with an N/A option
Fear of Hypoglycemia Survey (HFS-II) - Total Score, 2 Subscales and 4 Factor Scores | Screening, 13 weeks
  Fear of Hypoglycemia Survey (HFS-II) - total score, 2 subscales and 4 factor scores: Behavior (avoidance, maintain high BG), Worry (helplessness, social consequences)
The EuroQol 5 Dimension 5 Level (EQ-5D-5L) | Screening, 13 weeks
  The EQ-5D-5L is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical appraisal. The EQ-5D evaluates 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) using a 5-level severity scale from 1 (no problems) to 5 (extreme problems), and is converted to a single summary index by applying a formula that essentially attaches weight to each of the levels in each dimension. The visual analogue score (VAS) evaluates the health condition assessed by patients to producae a quantitive measure of health outcome that reflects the patient's own judgement on a range from "the worst health you can imagine" to "the best health you can imagine"
World Health Organization Well-being Index (WHO-5) | Screening, 13 weeks
  WHO-5 is a 5-item questionnaire of the World Health Organization that measures health related quality of life. Each item is scored on a scale of 0 (at no time) to 5 (all the time). Higher scores indicate greater well-being
Perceived Benefits and Burdens of AID Systems | Screening, 13 weeks
  A 35-item survey that assesses user expectations of a hybrid closed loop AID system using a 5-point Likert scale from "strongly disagree" to "strongly agree"
Total Daily Insulin (Units/kg) | 13 weeks
  Total daily insulin (Units/kg)
Percentage of Total Insulin Delivered Via Basal | 13 weeks
  Percentage of total insulin delivered via basal
Percentage of Total Insulin Delivered Via Bolus | 13 weeks
  Percentage of total insulin delivered via bolus
Weight | 13 weeks
  Weight
Body Mass Index (BMI) | 13 weeks
  Body Mass Index (BMI)
Number of Severe Hypoglycemia (SH) Events and SH Event Rate Per 100 person-years | 13 weeks
  Number of Severe Hypoglycemia (SH) events and SH event rate per 100 person-years
Number of Diabetes Ketoacidosis (DKA) Events and DKA Event Rate Per 100 person-years | 13 weeks
  Number of Diabetes Ketoacidosis (DKA) events and DKA event rate per 100 person-years
Number of Other Serious Adverse Events (SAEs other than SH events and DKA events) | 13 weeks
  Number of Other Serious Adverse Events (SAEs other than SH events and DKA events)
Number of Unanticipated Adverse Device Effects (UADE) | 13 weeks
  Number of Unanticipated Adverse Device Effects (UADE)
Number of Infusion Set Failures | 13 weeks
  Number of infusion set failures
Other Device Malfunctions/Device Issues | 13 weeks
  Number of other malfunctions/issues related to the study device

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Putman, MD, Study Chair — Massachusetts General Hospital; Colleen Bauza, PhD, MPH, Study Director — Jaeb Center for Health Research
Locations (16):
- United States (16):
  - University of Colorado-Barbara Davis Center for Diabetes, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Columbia University Medical Center, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia-Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No